CLINICAL TRIAL: NCT04965025
Title: MAGIC I TRIAL - Multi-stage Urethroplasty with Augmentation Using a Dorsal Graft Inlay Technique Comparing Graft Use in First or Second Stage: a Randomized Controlled Pilot Study
Brief Title: Multi-stage Urethroplasty with Augmentation Using a Dorsal Graft Inlay Technique Comparing Graft Use in First or Second Stage
Acronym: MAGIC I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-08585
Record Dates: First submitted 2020-09-30; First posted 2021-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urethra Stenosis; Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: RCT with two arms.
Masking Description: Participants cannot be blinded because of the nature of the surgery. Treating surgeon cannot be blinded. Blinding of outcome assessors, data analysts and authors of the manuscript was considered, but lifted due to practical considerations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-stage urethroplasty with graft inlay in first stage (Experimental)
  Interventions: Procedure: Multi-stage urethroplasty with graft inlay in first stage
- Multi-stage urethroplasty with graft inlay in second stage (Active Comparator)
  Interventions: Procedure: Multi-stage urethroplasty with graft inlay in second stage

INTERVENTIONS:
Procedure: Multi-stage urethroplasty with graft inlay in first stage — Herein, the graft will be used in the first stage and the second stage will solely consist of retubularizing the urethra.
  Arms: Multi-stage urethroplasty with graft inlay in first stage
Procedure: Multi-stage urethroplasty with graft inlay in second stage — Herein, the graft will be used in the second stage and the first stage will solely consist of opening the urethra longitudinally.
  Arms: Multi-stage urethroplasty with graft inlay in second stage

SUMMARY:
The principal aim of this pilot study is to directly compare both approaches and analyze the failure rate after one year of follow-up. These data will serve as the basis to design a larger phase II or III trial in the future with failure rate as the primary end-point. Other study objectives are thoroughly described underneath.

DETAILED DESCRIPTION:
Urethral stricture disease can occur throughout the entire length of the male urethra and has a wide variety of potential etiologies1. The standard treatment for this condition is urethroplasty, an open reconstructive procedure aiming to restore urethral patency1.

Urethroplasty covers a wide variety of surgical techniques and can be performed in a single stage or in multiple stages1. The latter option is generally reserved for patients with a very challenging disease1 (often including very dense fibrosis and poor local tissue conditions) and is most commonly performed for urethral strictures in the penile urethra2.

In case of a multi-stage urethroplasty, the first stage generally involves opening the urethra longitudinally over its diseased segment and suturing the urethral edges to the edges of the skin1. After that, a period of urethral rest of at least 3 months is foreseen after which the second stage procedure is performed by tubularizing the urethral plate around a transurethral catheter and closing the dartos layer and skin over the reconstructed urethra1. When the urethral plate is too narrow or of too poor quality to allow retubularization, the urethral plate is incised on the midline and a graft is sutured into the defect in order to augment the urethra enough to allow for retubularization after all1.

This dorsal inlay procedure can be performed during the first or second stage1. To the best of our knowledge, there are no studies that directly compare the outcomes of both approaches and consequently, there is no clear guidance for surgeons as to whether the graft should be administered during the first or second stage of the procedure. Also, there are absolutely no data available to use in a power analysis for a randomized controlled trial investigating this matter.

Against this background, the principal aim of this pilot study is to directly compare both approaches and analyze the failure rate after one year of follow-up. These data will serve as the basis to design a larger trial in the future with failure rate as the primary end-point. Other study objectives are thoroughly described underneath.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations.
* Age ≥ 18 years.
* Male patient.
* Fit for operation, upon surgeon's discretion.
* Isolated penile stricture that requires a multi-stage urethroplasty with dorsal inlay of a graft (upon surgeon's discretion).
* Use of oral mucosa as graft material.
* Patient is able and willing to comply with protocol.
* Prior urethral surgery (dilation, urethrotomy of urethroplasty) is allowed.

Exclusion Criteria:

* Absence of signed written informed consent.
* Age < 18 years.
* Female patients.
* Transgender patients.
* Patients unfit for operation.
* Stricture disease extending beyond the penile urethra or concomitant stricture at a different urethral segment.
* Use of graft other than oral mucosa.
* Any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study.
* Unwilling or unable to comply with study protocol.
* Patients deciding not to undergo the second stage will be excluded post-hoc.
* When the surgeon intra-operatively decides to carry out a single-stage procedure after all, the patient will also be excluded post-hoc.
* If the surgeon decides that no graft is needed to retubularize the urethra, the patient will also be excluded post-hoc.
* If the surgeon decides that a two-stage Bracka repair is needed, where the urethral plate is entirely cut away during the first stage and grafted, the patient will also be excluded post-hoc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To generate initial data in terms of failure rate after one year for grafting in first stage and for grafting in second stage. | After 1 year of follow-up after second stage
  * Failure will be defined as the inability to pass a 16 Fr flexible cystoscope through the reconstructed area without damaging the urethral mucosa.
  * A point-estimate with 95% confidence intervals will be made for the one year failure rate of grafting in first stage and grafting in second stage. These data will serve as the basis to design a larger trial in the future.

SECONDARY OUTCOMES:
To genarate initial data in terms of need for additional graft surgery for grafting in first stage. End-point time-frame: time period between first and second stage procedure. | 1 week after second stage surgery
  The absolute number and percentage of patients requiring additional graft surgery will be recorded.
  * Reasons for additional graft surgery will be recorded qualitatively.
  * Total number of grafts required will be recorded as well and will be presented as median with interquartile range for both treatment arms.
To generate initial data in terms of postoperative complications for grafting in first stage and for grafting in second stage. | Within 90 days after first stage and within 90 days after second stage.
  * Complications will be classified according to Clavien-Dindo4 and presented as absolute numbers with percentages for both treatment arms.
  * Types of complication will also be specified.
To generate initial data in terms of changes in erectile function for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  * International Index of Erectile Function (IIEF-5) questionnaire will be used (this is standard of care).
  * The IIEF-5 questionnaire provides a summative score between 5 and 25 and should be interpreted as follows: 22-25 = no erectile dysfunction; 17-21 = mild erectile dysfunction; 12-16 = mild to moderate erectile dysfunction; 8-11 = moderate erectile dysfunction; 5-7 = severe erectile dysfunction.
  * Change in erectile function at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To generate initial data in terms of changes in ejaculatory function for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  * Male Sexual Health Questionnaire - Ejaculatory Dysfunction short form (MSHQ-EjD) questionnaire will be used (this is standard of care).
  * The MSHQ-EjD short form questionnaire, consisting of 4 questions, provides a summative score between 1 and 15 (question 1 - 3) and a bother/satisfaction score between 0 and 5 (question 4).
  * Change in ejaculatory function at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To generate initial data in terms of changes in lower urinary tract symptoms for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  * International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms module (ICIQ-MLUTS) questionnaire and Peeling's voiding picture will be used (this is standard of care).
  * The ICIQ-MLUTS module, consisting of 7 questions, provides a summative score between 0 (asymptomatic) and 24 (most symptomatic) (question 1 - 6) and a bother score between 0 (not bothersome) and 3 (very bothersome) (question 7). Peeling's voiding picture provides a score between 1 and 4.
  * Change in lower urinary tract symptoms at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To generate initial data in terms of changes in urinary continence for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  * International Consultation on Incontinence Questionnaire - Urinary Incontinence short form (ICIQ-UI) questionnaire will be used (this is standard of care).
  * The ICIQ-UI short form questionnaire, consisting of 3 scoring questions and 1 self-diagnostic question, provides a summative score between 0 (asymptomatic) and 21 (most symptomatic).
  * Change in urinary continence at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To generate initial data in terms of changes in quality of life for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  * The 3-level version of the EQ-5D (EQ-5D-3L) questionnaire and the EQ Visual Analogue Scale (EQ-VAS) will be used (this is standard of care).
  * The EQ-5D-3L questionnaire, consisting of 5 questions, provides a 5-digit score in which every digit varies between 1, 2 and 3. The EQ-VAS provides a scale between 0 and 100.
  * Change in quality of life at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To generate initial data in terms of (changes in) patient satisfaction for grafting in first stage and for grafting in second stage. | 3 months after second stage and 1 year after second stage.
  * Two specific questions about patient satisfaction will be used (this is standard of care).
  * The results of these two questions will be presented as absolute numbers with percentages for each possible answer for both treatment arms.
To generate initial data in terms of change in maximal urinary flow rate (Qmax) for grafting in first stage and for grafting in second stage. | Preoperative, 3 months after first stage (before second stage), 3 months after second stage and 1 year after second stage.
  - Change in Qmax at the aforementioned moments will be presented as median change in score compared to baseline with interquartile range for both treatment arms.
To assess feasibility of randomization. | After 12 motnhs of follow-up
  * The proportion of patients randomized over all patients undergoing multi-stage urethroplasty with dorsal inlay of a graft that were screened for the trial will be used to assess feasibility.
  * A proportion of 0.70 or higher will be considered as 'feasible'.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, Principal Investigator — University Hospital, Ghent; Wesley Verla, Study Director — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request only